CLINICAL TRIAL: NCT03015831
Title: Effect of Low Dose ColchiciNe on the InciDence of Atrial Fibrillation in Open Heart Surgery Patients
Brief Title: Effect of Low Dose ColchiciNe on the InciDence of POAF
Acronym: END-AFLD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Statistical analysis of interim data showed no advantage of colchicine
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JordanCCG
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation; Cardiac Surgery; Colchicine Adverse Reaction
Keywords: Atrial fibrillation; Cardiac surgery; Colchicine
MeSH Terms: conditions — Atrial Fibrillation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Active Comparator): Intervention by administering an active copmarator of 1 mg colchicine one day pre op and 0.5 mg daily after surgery until discharge
  Interventions: Drug: Colchicine
- Placebo Oral Tablet (Placebo Comparator): Identical tablet (placebo) administered in a similar way as that in the active comparator arm
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Colchicine — Colchicine will be given to open heart surgery patients
  Other Names: Colcrys, Mitigare
  Arms: Colchicine
Drug: Placebo Oral Tablet — Placebo Oral Tablet will be given to open heart surgery patients according to randomization
  Other Names: Placebo
  Arms: Placebo Oral Tablet

SUMMARY:
The prior End-AF study by the same group showed that 1 mg of colchicine didn't decrease the incidence of AF after cardiac surgery. The current study, End-AF Low Dose Study, will test 0.5 mg colchicine vs. placebo in preventing AF after cardiac surgery.

DETAILED DESCRIPTION:
AF after cardiac surgery leads to excess mortality and morbidity. Colchicine was used in several studies to lower the incidence AF but the results were generally disappointing. There was no benefit in reducing AF and there was a high incidence of GI side effects especially diarrhea, often leading to stopping the medication. However, a recently published meta-analysis showed that colchicine reduced AF, but again warned of the high incidence of GI side effects. The maintenance dose of colchicine used in these studies was 1 mg daily it is hypothesized that low dose colchicine (0.5 not 1 mg colchicine) might lower AF after cardiac surgery without the prohibitive GI side effects Patients will be randomized to colchicine vs. placebo started the day before surgery and continued until hospital discharge.

The primary efficacy endpoint will be the incidence of AF. The primary safety endpoint will be the GI side effects

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or above undergoing elective cardiac surgery.
* Sinus rhythm and no previous AF
* Agreed to sign informed consent.

Exclusion Criteria:

* Known severe liver disease or current transaminases >1.5 times the upper normal limit
* Current serum creatinine >2.5 mg/dL
* Known myopathy or elevated baseline preoperative creatine kinase
* Known blood dyscrasias or significant gastrointestinal disease
* Pregnant and lactating women
* Known hypersensitivity to colchicine
* Current treatment with colchicine for any indications
* Emergency surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | Through study completion, an average of 1 week
  AF documented by EKG

SECONDARY OUTCOMES:
Side effects of colchicine | Through study completion, an average of 1 week
  Gastrointestinal side effects

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Tabbalat, MD, FACC, Principal Investigator — JCC Group, Cardiology Department, Khalidi Medical Center, Amman, Jordan
Locations (3):
- Jordan (3):
  - Istishari Hospital, Amman
  - Jordan Hospital, Amman
  - Khalidi Hospital & Medical Center, Amman

IPD SHARING:
Plan to Share IPD: Yes
Our Group's website will share data. Researchgate will share data. Eventual results will be announced to medical community through local presentations, and international congresses and publications.

REFERENCES:
- [Derived] Tabbalat RA, Alhaddad I, Hammoudeh A, Khader YS, Khalaf HA, Obaidat M, Barakat J. Effect of Low-dose ColchiciNe on the InciDence of Atrial Fibrillation in Open Heart Surgery Patients: END-AF Low Dose Trial. J Int Med Res. 2020 Jul;48(7):300060520939832. doi: 10.1177/0300060520939832. PMID 32720823